CLINICAL TRIAL: NCT06059547
Title: A Multi-center Phase 2 Study of Neoadjuvant Immunotherapy in Combination With the Anti-GDF-15 Antibody Visugromab (CTL-002) for the Treatment of Muscle Invasive Bladder Cancer
Brief Title: Neoadjuvant Immunotherapy Combined With the Anti-GDF-15 Antibody Visugromab to Treat Muscle Invasive Bladder Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CatalYm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTL-002-002
Record Dates: First submitted 2023-08-23; First posted 2023-09-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer; Adult Solid Tumor
Keywords: CTL-002; visugromab; GDF-15
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Participants will be stratified into four cohorts based on disease stage and PD-L1 expression. Within each cohort, participants are centrally and sequentially assigned to one of two treatment arms in a non-randomized, parallel assignment model.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination with Placebo (Active Comparator): Placebo + Checkpoint Inhibitor nivolumab
  Interventions: Drug: Nivolumab; Drug: Placebo
- Combination with Visugromab/Verum (Experimental): visugromab (CTL-002) + Checkpoint Inhibitor nivolumab
  Interventions: Drug: Nivolumab; Drug: Visugromab (CTL-002)

INTERVENTIONS:
Drug: Nivolumab — Biological, monoclonal antibody
Drug: Visugromab (CTL-002) — Biological, monoclonal antibody
  Arms: Combination with Visugromab/Verum
Drug: Placebo — Placebo (NaCl) for Visugromab (CTL-002)
  Arms: Combination with Placebo

SUMMARY:
This is a multi-center, stratified and single-blinded Phase 2 trial of neoadjuvant immunotherapy in combination with the anti-GDF15 antibody visugromab (CTL-002) for the treatment of participants with MIBC set to undergo radical Cystectomy (RC)/Re-TURBT who cannot receive or refuse to receive cisplatin-based chemotherapy.

ELIGIBILITY:
Main Inclusion Criteria:

* Signed and dated informed consent, and able to comply with the study procedures and any locally required authorization.
* Male or female aged ≥ 18 years.
* Histopathologically confirmed urothelial carcinoma.
* Clinical Stage T2-T4aN0M0 MIBC.
* Ineligible for cisplatin therapy per modified Galsky criteria or refuses cisplatin-based chemotherapy.
* Eligible for radical Cystectomy.
* Pretreatment tumor material from transurethral resection of the bladder tumor (TURBT) must be available.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Adequate organ function (bone marrow, hepatic, renal function and coagulation).

Main Exclusion Criteria:

* Pregnant or breastfeeding.
* Received prior radiotherapy on the bladder tumor.
* Received a partial cystectomy.
* Any prior systemic anti-cancer therapy including investigational agents and immunotherapy.
* Following cardio-vascular risk factors:

  1. Myocardial infarction in the past 6 months before planned treatment start.
  2. Uncontrolled heart failure.
  3. Uncontrolled ventricular arrhythmia.
  4. A peri/myocarditis in the past 3 months before planned treatment start. Note: Stable atrial fibrillation is permissive with or without anticoagulation if there was no decompensation in the past 3 months before planned treatment start.
* Left ventricular ejection fraction (LVEF) < 50% measured by echocardiogram or MUGA.
* QTcF ≥ 470 ms regardless of sex.
* Any active autoimmune requiring systemic immunosuppressive treatments.
* Any history of non-infectious pneumonitis < 6 months prior to Screening.
* Any active inflammatory bowel disease such as Crohn's disease or ulcerative colitis which are generally excluded or active autoimmunthyroiditis present < 6 months prior to Screening.
* History of CNS disease such as stroke, seizure, encephalitis, or multiple sclerosis (< 6 months prior to Screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | min. 4 months
  Rate of participants with complete pathological responses after IMP treatment as determined by local pathologist review
Radiological response rate according RECIST | min. 4 months
  Rate of participants with radiological responses according to RECIST 1.1 prior Radical Cystectomy/Re-TURBT as assessed by the Investigator/Radiologist

SECONDARY OUTCOMES:
Adverse Events | min. 6 months
  Incidence of adverse events (related or unrelated to IMPs)
Treatment related delay of surgery | min. 6 months
  Treatment related delay of Radical Cystectomy/Re-TURBT > 8 weeks after last dose of IMP
Cmax following the first dose of Visugromab (CTL-002) | 1 day
  PK parameter from serum Visugromab (CTL-002) levels
AUC following the first dose of Visugromab (CTL-002) | 28 days
  PK parameter from serum Visugromab (CTL-002) levels
Half-life of Visugromab (CTL-002) | min. 3 months
  PK parameter from serum Visugromab (CTL-002) levels
GDF-15 serum levels | 1 day
  Measurement of concentration in peripheral blood
Pathological complete response rate | min. 4 months
  Rate of participants with complete pathological responses after IMP treatment as determined by central independent pathological review
Radiological response rate according RECIST | Min. 4 months
  Rate of participants with radiological responses according to RECIST 1.1 prior Radical Cystectomy/Re-TURBT as assessed by the central independent review
Major pathological response rate | Min. 4 months
  Rate of participants with major pathological responses after IMP treatment as determined by local pathologist review or central independent pathological review
Evaluation of EFS (Event-free Survival) | 12 months after Radical Cystectomy/Re-TURBT
  Event-free survival will be defined as the time from first IMP administration to one of the following:
  Radiographic disease progression precluding a curative intent surgery per RECIST v1.1 prior to RC/Re-TURBT.
  Initiation of neoadjuvant chemotherapy preceding RC/Re-TURBT as per Investigator decision.
  Inability to undergo RC/Re-TURBT due to the onset of treatment-related side effects.
  Inability to complete a curative intent surgery determined by the urologist at the time of RC/Re-TURBT (e.g., unresectable tumor, metastases discovered at RC).
  Local or distant recurrence assessed by cross-sectional imaging and/or biopsy after RC/Re-TURBT.
  Death from any cause. In this trial, participant refusal to undergo RC due to the evidence of complete or near-complete clinical response (assessed on cross-sectional imaging as previously described) will not be considered an event.
OS (Overall Survival) | 15 months
  Overall survival is defined as the time from the first IMP administration to the date of death, regardless of the cause of death.
  Participants who were alive at the time of the analysis will be censored at the date the participant was last known to be alive.
Evaluation of TTR (Time to Relapse) | 12 months after Radical Cystectomy/Re-TURBT
  Time to relapse will be measured from the time of RC/Re-TURBT until the day of documented relapse.
Visugromab-induced anti-drug antibodies (ADA) development. | min. 5 months
  The number and percentage of participants with any detectable ADA after first IMP administration

OTHER OUTCOMES:
Tumor biopsy analysis | min. 3 months
Evaluation of selected cytokine and chemokine concentration in peripheral blood | min. 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Felix Lichtenegger, MD, Study Director — CatalYm GmbH
Locations (4):
- Italy (4):
  - IRCCS Ospedale San Raffaele Hospital Vita-Salute San Raffaele University, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, UOC Oncologia Medica, Roma
  - A.O.U. Città della Salute e della Scienza di Torino, Torino

IPD SHARING:
Plan to Share IPD: No